CLINICAL TRIAL: NCT01099332
Title: CopperProof-2: Prospective, Randomized, Double-Blind Placebo-Controlled Clinical Trial Comparing the Effects of a Novel Once-Daily Oral Zinc Cysteine Preparation on Zinc and Copper Parameters in Mild Cognitive Impairment and Alzheimer's Disease
Brief Title: Trial of Novel Oral Zinc Cysteine Preparation in Alzheimer's Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Adeona Pharmaceuticals (Industry)
Responsible Party: Diana Pollock, M.D., P.I., Neurology Research Unit of Clearwater FL
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CopperProof-2
Record Dates: First submitted 2010-03-30; First posted 2010-04-07 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
Keywords: Alzheimer's disease; Mild Cognitive Impairment; Copper metabolism; Zinc metabolism; Ceruloplasmin
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gastro-retentive zinc cysteine tablet (Active Comparator): Once daily administration by mouth of a gastro-retentive, sustained-release preparation of zinc cysteine with excipients, all G.R.A.S., with adequate water.
  Interventions: Other: Gastro-retentive zinc cysteine tablet
- Identical appearance of placebo with active comparator (Placebo Comparator): Once daily administration of placebo of identical physical appearance to that of active comparator with similar amount of water.
  Interventions: Other: Tablet identical physically to active comparator containing some lactose

INTERVENTIONS:
Other: Gastro-retentive zinc cysteine tablet — Oral, one tablet, once daily with water for 6 months.
  Other Names: Zinthionein ZC
  Arms: Gastro-retentive zinc cysteine tablet
Other: Tablet identical physically to active comparator containing some lactose — Oral, once daily, with water, 6 months.
  Other Names: Placebo Tablet
  Arms: Identical appearance of placebo with active comparator

SUMMARY:
This trial aims to test the hypothesis that 1) a single dose of zinc cysteine in a proprietary gastro-retentive form will produce sustained blood levels of zinc giving a larger bioavailable amount of zinc than an FDA approved preparation of inorganic zinc acetate; and 2) that the zinc cysteine gastro-retentive, sustained-release preparation will be better tolerated with significantly less gastrointestinal side effects than the zinc acetate capsules. The trial also tests the hypothesis that, after 6 months of once daily administration, the zinc cysteine subjects will show reduced serum non-ceruloplasmin copper. Additionally, subjects will perform tests of mental function,including the dementia rating scale, the Mini Mental Status Examination and the ADAS-cognitive performance test aimed at Alzheimer's status assessment. Tests will be administered at baseline, 3 and 6 months, and the performance results compared. Care-giver assessments will also be noted.

DETAILED DESCRIPTION:
This multi-center study aims to determine the pharmacokinetics and pharmacodynamics of a novel gastro-retentive, sustained-release zinc cysteine preparation on the blood and urine measures of copper and zinc balance in Alzheimer's disease and mild cognitive impairment. Data expected to be derived include tolerability of the novel preparation in comparison with oral inorganic zinc salt, and long-term effects on primarily blood-measured copper-zinc balance. The study design is that of a prospective, randomized, double blind placebo-controlled clinical trial, with a duration for individual subjects of 6 months. The study will be performed at a total of 3 sites, under the direction of a single principal investigator, with a sub-investigator. The statistical plan calls for a comparison of data from the two long-term parallel groups using ANOVA and other applicable techniques. In addition to blood parameters, mental function assessments obtained at baseline, 3 and 6 months will be evaluated statistically.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's disease mild to moderate as diagnosed by standard clinical, functional and NINDA-ADRDA criteria
* Mild cognitive impairment diagnosed by standard clinical, functional and NINDA-ADRDA criteria
* All subjects able to swallow Tablets
* Subjects taking copper or zinc containing supplements must have a 30-day wash out before starting study materials
* Screening laboratory values either within normal limits or deemed not clinically significant by investigator

Exclusion Criteria:

* Subjects or their study companions/care givers unable to give adequate informed consent
* Presence of a disease or condition known to affect biometal homeostasis
* Presence of psychosis, substance abuse or other major medical or neurological issues
* Presence of vascular dementia
* Clinically significant anemia at the time of the screening visit
* Current use of a decoppering drug such as trientine or penicillamine

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Biometal levels will be measured in serum by atomic absorption spectrometry | 6 to 12 months
  Active comparator material orally administered will be associated with better tolerability than oral zinc acetate, and will produce a reduction in serum non-ceruloplasmin bound copper levels and an elevation in serum zinc levels

SECONDARY OUTCOMES:
Serum zinc levels after oral administration of two different zinc-containing compounds and placebo will be determined by atomic absorption spectrometry | 3 months
  The change in serum zinc levels over time after oral administration of the active comparator of the study as well as the placebo and for certain subjects an inorganic zinc salt will be compared
Comparison of mental status functions at baseline, 3 and 6 months in active comparator versus placebo groups. | 6 to 12 months
  All subjects will perform standard and standardized tests of mental function, ranging from a general dementia rating scale (Mini Mental Status Exam) to more Alzheimer's specific tests (ADAS-cognitive). Daily living and caregiver assessments of overall daily functioning will be noted. Test results will be compared statistically in a two-point fashion, and correlated with biometal ststus.

CONTACTS AND LOCATIONS:
Overall Officials: David Newsome, M.D., Study Director — Senior Vice President of Research and Development, Adeona Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Neuroscience Research Unit, Clearwater, Florida
  - ATIT Neurology, Holiday, Florida
  - The Cottages, Port Richey, Florida

REFERENCES:
- [Background] Squitti R, Bressi F, Pasqualetti P, Bonomini C, Ghidoni R, Binetti G, Cassetta E, Moffa F, Ventriglia M, Vernieri F, Rossini PM. Longitudinal prognostic value of serum "free" copper in patients with Alzheimer disease. Neurology. 2009 Jan 6;72(1):50-5. doi: 10.1212/01.wnl.0000338568.28960.3f. PMID 19122030
- [Background] Arnal N, Cristalli DO, de Alaniz MJ, Marra CA. Clinical utility of copper, ceruloplasmin, and metallothionein plasma determinations in human neurodegenerative patients and their first-degree relatives. Brain Res. 2010 Mar 10;1319:118-30. doi: 10.1016/j.brainres.2009.11.085. Epub 2009 Dec 22. PMID 20026314
- [Background] Brewer GJ, Newsome DA et al. Sub-clinical zinc deficiency found in Alzheimer's disease. Presented at ICAD, Vienna,Austria; July 2009 09-HT-2656-ALZ; submitted for publication